CLINICAL TRIAL: NCT01976546
Title: Intubation With McGrath Video Laryngoscope and Boedeker Intubation Foreceps in a Population of Patients With Predictors of Difficult Airway, an Observational Pilot Study
Brief Title: Intubation With McGrath Video Laryngoscope and Boedeker Intubation Foreceps in a Population of Patients With Predictors of Difficult Airway
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Camilla Strøm, M.D, Rigshospitalet, Denmark
Other Study IDs: LP-CS-13
Record Dates: First submitted 2013-10-29; First posted 2013-11-06 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Patients With One or More Predictors of Difficult Airway
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- airway: Patients with one or more predictors of diffucult airway
  Interventions: Device: Intubation with mcgrath videolaryngoscope and Boedeker intubation foreceps

INTERVENTIONS:
Device: Intubation with mcgrath videolaryngoscope and Boedeker intubation foreceps — Patients will be intubated with the Mcgrath videolaryngoscope and a tracheal tube placed by Boedeker intubation foreceps
  Other Names: Aircraft Medical McGRATH series 5 videolaryngoscope; Karl Storz Boedeker intubation foreceps

SUMMARY:
Tracheal intubation with videolaryngoscopes have been widely studied, and is now often used in the management of difficult airways.

Videolaryngoscopes with angulated blades can improve laryngeal view, however this does not always match with a higher intubation succes. To adress this matter the aim of this study is gathering experience with intubation with mcgrath videolaryngoscope and a blade-shape intubation foreceps (Boedeker intubation foreceps, Karl Storz, Germany).

The hypothesis is that intubation with this combination is easy and can be a good alternative when using the McGrath videolaryngoscope in patients with predictors of difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective surgery
* age over 18 or more
* planned intubation with mcgrath videolaryngoscope
* informed conscent obtained
* patients are
* patients shall be able to read and understand Danish

Exclusion Criteria:

* Patients planned to awake intubation
* stridor
* hypoxia defined by saturation under 90% without oxygen supply
* patients with oxygentreatment at home
* patients that need a wired tube
* patients that need a preshaped tube
* patients that need crash induction
* use of gastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with one or more predictors of difficult airway
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to intubation | within one day

SECONDARY OUTCOMES:
Sore throat | within 2 days
succesful intubation | within one day
Damage on teeth | 2 days
Intubation difficulty | within one day
  Intubation difficulty scale
Intubation conditions | within one day
  a.m fuchs-buder
Intubation attempts | within one day

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Strøm, M.D, Principal Investigator — Dept. of anaesthesia, centre of head and orthopedics, Rigshospitalet, Denmark
Locations (1):
- Dept. of Anaesthesia, Centre of Head and Orthopedics 4231, Rigshospitalet, Copenhagen, Denmark